CLINICAL TRIAL: NCT01766089
Title: Comparison Between Dexmedetomidine and Remifentanil on the Maternal Responses to Tracheal Intubation in Severe Pre-eclamptic Patients During Caesarean Delivery
Brief Title: Dexmedetomidine vs. Remifentanil for Pre-eclampsia During Caesarean Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R/61; R/61 (Other Grant/Funding Number: Mansoura University, Mansoura, Egypt)
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy; Severe Pre-eclampsia
Keywords: Caesarean delivery; severe pre-eclampsia; remifentanil; dexmedetomidine; cardiovascular response
MeSH Terms: conditions — Pre-Eclampsia | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): dexmedetomidine intravenous infusion rate of 0.4 µg/kg/h
  Interventions: Drug: Dexmedetomidine
- Remifentanil (Placebo Comparator): remifentanil intravenous infusion rate of 0.1 µg/kg/min
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil (0.1 µg/kg/min) starting 5 min before induction of anaesthesia and continued until peritoneal closure.
  Arms: Remifentanil
Drug: Dexmedetomidine — dexmedetomidine (0.4 µg/kg/h) starting 20 before induction of anaesthesia and continued until peritoneal closure
  Arms: Dexmedetomidine

SUMMARY:
Preeclampsia is a pregnancy-specific, multisystem disorder that complicates approximately 5 % of pregnancies.

Tracheal intubation in the women with severe pre-eclampsia is usually associated with exaggerated transient increases in blood pressure, heart rate and maternal plasma catecholamine concentrations. These changes may lead to maternal cerebral oedema, haemorrhage, left ventricular failure, pulmonary oedema or mortality, and reduce uterine blood flow which may adversely affect the neonatal wellbeing. Therefore, the attenuation of the haemodynamic responses to tracheal intubation in this unique group of patients is demanding for the best of both mother and foetus.

The use of single remifentanil boluses of 0.5 to 1 µg/kg reduces effectively the haemodynamic and catecholamine responses to laryngoscopy and tracheal intubation in severe pre-eclamptics during Cesarean delivery under general anesthesia. Unfortunately, the use of 1 µg/kg doses are associated with more maternal hypotension and neonatal respiratory depression requiring resuscitation. Moreover, the use of preinduction remifentanil bolus of 0.5 µg/kg followed by a continuous infusion at 0.15-0.2 µg/kg/min is associated with significant attenuation of the maternal stress response to tracheal intubation with variable degree of neonatal depression in non-pre-eclamptic women. Whereas, the use of infusion rates of 0.1 µg/kg/min or less is less likely to produce neonatal depression.

In our previous study, we demonstrated that the preoperative administration of dexmedetomidine 0.4 and 0.6 µg/kg/h, a specific alpha 2-adrenoceptor agonist, blunts the maternal haemodynamic and hormonal responses to Caesarean delivery under sevoflurane anaesthesia without adverse neonatal effects. However the use of 0.6 µg/kg/h doses is associated with higher postoperative sedation scores.

DETAILED DESCRIPTION:
We hypothesize that the preoperative intravenous dexmedetomidine (0.4 µg/kg/h) and remifentanil (0.1 µg/kg/min) infusions will have comparable maternal haemodynamic responses to tracheal intubation, surgical stimulation and extubation after uncomplicated Caesarean delivery under general anesthesia in parturients with severe pre-eclampsia, without adverse neonatal effects.

Anaesthetic management will be standardized in all studied patients. Oral ranitidine 150 mg and metoclopramide 10 mg will be given the night before and on the morning of surgery, with 0.3 mol/L sodium citrate 30 mL given 15 min before induction. Magnesium sulphate will be given as a loading dose of 4 g intravenously, followed by i.v. infusion of 1g/hour for seizures prophylaxis.

Intravenous boluses of hydralazine 5 mg at 20-min intervals will be used if SAP increases above 160 mm Hg or DAP above 110 mm Hg, to keep the diastolic blood pressure at approximately 90 mmHg and the doses used will be recorded.

The studied population will be allocated randomly to one of two groups, (n = 18, in each), by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomization code (Random Allocation Software, version 1.0.0, Isfahan University of Medical Sciences, Isfahan, Iran), to receive either dexmedetomidine (0.4 µg/kg/h) or remifentanil (0.1 µg/kg/min) starting 20 and 5 min before induction of anaesthesia, respectively, and will be discontinued after peritoneal closure. The dexmedetomidine and remifentanil solutions looked identical.

One anaesthesiologist who is not otherwise involved in the study, will prepare the study solutions, install them in the infusion pumps, set up the dose according to the assigned randomized dose, and will mask the infusion pumps with an opaque sheet throughout the procedure to ensure the blindness of the assessors. Another anaesthesiologist who will be blinded to treatment regimen provided perioperative care. A third anaesthesiologist will collect perioperative data. All staff in the operating room will be unaware of patient allocation.

Maternal monitoring will include three lead-electrocardiography, non-invasive blood pressure, and pulse oximetry. Left uterine displacement will be maintained.

After preoxygenation for 3 min, rapid sequence induction will be performed using propofol 1.5-2.5 mg/kg and suxamethonium 1 mg/kg with the application of cricoid pressure from the time of loss of the consciousness until the inflation of the cuff of the endotracheal tube. Laryngoscopy will be performed after the 1-min blood pressure recording, and tracheal intubation will be completed before the 2-min reading. Correct placement of the endotracheal tube will be confirmed with direct visualization of the passage of its tip between the vocal cords, auscultation of equal breath sounds on both sides of the chest and capnography waveform. The patient's lungs will be mechanically ventilated to maintain (ETCO2) at 30-35mmHg. Anaesthesia will be maintained with a 0.5-0.7% minimum alveolar concentration of sevoflurane in oxygen. Atracurium 0.5 mg/kg will be given for muscle relaxation to maintain suppression of the second twitch using a train-of-four stimulation. The Induction-to-delivery time will be recorded using a stopwatch.

After the umbilical cord is clamped, a 5-10 IU infusion of oxytocin in 500 mL of lactated Ringer's solution will be started and morphine 0.1 mg/kg will be given. After peritoneal closure, study solution will be discontinued.At the end of surgery, sevoflurane will be discontinued, residual neuromuscular block will be antagonized and the trachea will be extubated.

Postoperative analgesia will be achieved according to the authors' hospital protocol with 12-hourly IM diclofenac (75 mg), 6-hourly IVI paracetamol (1 g), and rescue doses of IV meperidine (25 mg).

Statistical analysis:

Data will be tested for normality using the Kolmogorov-Smirnov test. X2 test will be used for categorical data. Repeated-measures analysis of variance will be done to test the serial changes in hemodynamic and cortisol data. Student-t- and Mann Whitney U tests will be used to compare the parametric and nonparametric data between the two studied groups. Data will be expressed as mean (SD), number (%), or median [range]. p < 0.05 will be considered to represent statistical significance.

In a previous study, Yoo et al have demonstrated that the mean (SD) values of MAP at 1 min after tracheal intubation in those received remifentanil bolus were 118 (20) mm Hg. A priori power analysis revealed that 16 patients would be needed in each group to detect a 20% difference in MAP values, 1 min after intubation, after the administration of remifentanil with a type I error of 0.05 and a power of 90%. We assumed that the detection of 20% differences in the mean MAP would be of clinically importance. We increased the sample size by 10% to compensate for patients dropping out during the study.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 34 weeks
* severe pre-eclampsia
* symptoms of imminent eclampsia
* Caesarean delivery
* General anaesthesia

Exclusion Criteria:

* allergy to dexmedetomidine
* cardiac disease
* pulmonary disease
* hepatic disease
* renal disease
* neurological disease
* neuromuscular disease
* body mass index >35kg/m2
* diabetes mellitus
* anemia
* coagulation disorders
* bleeding disorders
* seizures
* Hemolysis, Elevated Liver enzymes and Low platelet count (HELLP) syndrome
* receiving cardiovascular medications
* receiving antipsychotic medications
* receiving hypnotic medications
* alcoholic
* drug abuse
* foetal distress
* placenta praevia
* abruptio placenta
* multiple pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure | Changes from baseline for 60 min after delivery
  Mean blood pressure

SECONDARY OUTCOMES:
Systolic blood pressure | Changes from baseline for 60 min after delivery
  Systolic blood pressure
Heart rate | Changes from baseline for 60 min after delivery
  Heart rate
Diastolic blood pressure | Changes from baseline for 60 min after delivery
  Diastolic blood pressure
neonatal Apgar scores | from delivery to 5 minutes after that
  Apgar scores
Neurologic and adaptive capacity score | for 24 hours after delivery
  Neonatal neurologic and adaptive capacity score (NACS)
Maternal Cortisol | from baseline for 1 hour after delivery
  Plasma cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Samah El Kenany S, MD, Study Chair — Lecurer of Anesthesiology; Eyad A Ramzy, MD, Study Chair — Lecturer of Anesthesiology and Pain Management; Ehsan M Abdelaty, MD, Study Chair — Lecturer of Clinical Pathology
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt